CLINICAL TRIAL: NCT02107014
Title: Low Dose Naltrexone (LDN) Immune Monitoring
Acronym: LDN-IM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Stanford University (Other)
Responsible Party: Principal Investigator, Jarred W. Younger, Associate Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 29911
Record Dates: First submitted 2014-04-01; First posted 2014-04-08 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-02

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Low Dose Naltrexone (LDN) (Other): Following a two-week baseline the study drug was administered daily for 8 weeks. Participants were informed that placebo or LDN would be provided during the drug period and that all participants would receive LDN at some point during the study. In fact, all participants received the active LDN (4.5 mg nocte) throughout the drug-administration period.
  Interventions: Drug: Low Dose Naltrexone

INTERVENTIONS:
Drug: Low Dose Naltrexone — Naltrexone 4.5 mg p.o. nocte
  Other Names: LDN; Naltrexone

SUMMARY:
We have found that low dose naltrexone (LDN) can substantially reduce pain associated with fibromyalgia syndrome. We believe LDN may work via novel anti-inflammatory channels. The purpose of this study is to determine if LDN lowers inflammatory markers in individuals with fibromyalgia.

DETAILED DESCRIPTION:
Eligible women with Fibromyalgia (FM) will be enrolled into a 10-week drug trial. During the first two weeks, a baseline phase will be used to collect data on immune function and symptoms. LDN will be administered for 8 weeks. Although there is no placebo arm built-in, participants will be advised that they may receive a placebo during the trial. Participants will provide twice daily symptom reports using an android tablet device and Dooblo SurveyToGo survey software. Participants will also provide a blood sample twice every week for the duration of the study. Plasma inflammatory markers will be tested using a luminex based 63-plex inflammatory assay panel.

The primary aim of the study is to test if 8 weeks of LDN administration is associated with a reduction in pro-inflammatory markers in plasma in women with FM.

ELIGIBILITY:
Inclusion Criteria:

* Females age 18-65
* Meets criteria for 1990 ACR criteria for fibromyalgia
* Able to receive venous blood draw twice a week for 16 weeks
* Sufficient symptom variability during baseline report
* Patient completes daily report during 2 week baseline period at least 80% completion rate.

Exclusion Criteria:

* Opioid use
* Significant psychological comorbidity that in the discretion of the investigator compromises study integrity
* Location prohibits travel to Stanford
* Blood or clotting disorder
* Rheumatologic or autoimmune disease
* Acute infection
* Baseline blood ESR >60, CRP greater than 3.0mg/L, positive rheumatoid factor, or positive ANA
* Use of blood thinning medication
* Pregnant or currently planning to become pregnant
* Current use of aspirin, ibuprofen, naproxen, or other confounding-anti-inflammatory medication as part of regular medication regimen.
* Known allergy to Naltrexone or Naloxone
* Currently participating in another treatment-based research study
* Self-reported inability to refrain from alcohol for the duration of the study period

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jarred Younger, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Stanford University School of Medicine, Palo Alto, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited Feb-April 2014 from a laboratory database of individuals with fibromyalgia who are interested in participating in research.
Period: Overall Study
Arm/Group | Low Dose Naltrexone (LDN)
Started | 9
Completed | 8
Not Completed | 1
Not completed — Withdrew before drug: moving interstate | 1

BASELINE CHARACTERISTICS:
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in IL-1α From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  IL-1α baseline 2-weeks | 3.56 [3.52 to 4.43]
  IL-1α last 2-weeks | 3.88 [3.79 to 4.74]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = .576, Mixed Models Analysis

2. Primary Outcome: Change in IL-1β From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  IL-1β baseline 2-weeks | 0.33 [0.16 to 14.98]
  IL-1β last 2-weeks | 0.26 [.04 to 10.88]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.010, Mixed Models Analysis

3. Primary Outcome: Change in IL-1Ra From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  IL-1Ra baseline 2-weeks | 2433.11 [2406.25 to 2500.26]
  IL-1Ra last 2-weeks | 2004.48 [1846.09 to 2164.39]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = .008, Mixed Models Analysis

4. Primary Outcome: Change in IL-2 From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  IL-2 baseline 2-weeks | 23.21 [4.98 to 105.98]
  IL-2 last 2-weeks | 21.32 [4.98 to 83.43]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = .015, Mixed Models Analysis

5. Primary Outcome: Change in IL-4 From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  IL-4 baseline 2-weeks | 20.70 [14.63 to 100.50]
  IL-4 last 2-weeks | 19.00 [13.10 to 83.48]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = .007, Mixed Models Analysis

6. Primary Outcome: Change in IL-5 From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  IL-5 baseline 2-weeks | 1.94 [1.33 to 18.46]
  IL-5 last 2-weeks | 4.57 [1.24 to 11.28]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = .016, Mixed Models Analysis

7. Primary Outcome: Change in IL-6 From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  IL-6 baseline 2-weeks | 10.22 [9.46 to 27.85]
  IL-6 last 2-weeks | 5.87 [3.64 to 23.27]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p < 0.001, Mixed Models Analysis

8. Primary Outcome: Change in IL-7 From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  IL-7 baseline 2-weeks | 10.18 [9.31 to 16.34]
  IL-7 last 2-weeks | 10.28 [8.31 to 14.99]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.212, Mixed Models Analysis

9. Primary Outcome: Change in IL-8 From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  IL-8 baseline 2-weeks | 0 [0 to 0]
  IL-8 last 2-weeks | 0 [0 to 0]

10. Primary Outcome: Change in IL-9 From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  IL-9 baseline 2-weeks | 0 [0 to 0]
  IL-9 last 2-weeks | 0 [0 to 0]

11. Primary Outcome: Change in IL-10 From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  IL-10 baseline 2-weeks | 6.01 [5.26 to 67.43]
  IL-10 last 2-weeks | 10.11 [6.35 to 52.87]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.008, Mixed Models Analysis

12. Primary Outcome: Change in IL-12p40 From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  IL-12p40 baseline 2-weeks | 6.91 [4.74 to 11.12]
  IL-12p40 last 2-weeks | 6.43 [5.09 to 9.76]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.004, Mixed Models Analysis

13. Primary Outcome: Change in IL-12p70 From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  IL-12p70 baseline 2-weeks | 1.82 [1.68 to 6.28]
  IL-12p70 last 2-weeks | 1.69 [1.60 to 5.47]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p < 0.001, Mixed Models Analysis

14. Primary Outcome: Change in IL-13 From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  IL-13 baseline 2-weeks | 0.66 [0.16 to 8.58]
  IL-13 last 2-weeks | 0.66 [0.31 to 7.21]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.047, Mixed Models Analysis

15. Primary Outcome: Change in IL-15 From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  IL-15 baseline 2-weeks | 11.08 [7.07 to 119.95]
  IL-15 last 2-weeks | 8.71 [7.07 to 105.88]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.002, Mixed Models Analysis

16. Primary Outcome: Change in IL-17A From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  IL-17A baseline 2-weeks | 5.03 [3.05 to 26.86]
  IL-17A last 2-weeks | 3.40 [2.05 to 24.02]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.003, Mixed Models Analysis

17. Primary Outcome: Change in IL-17F From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  IL-17F baseline 2-weeks | 0.95 [0.80 to 12.02]
  IL-17F last 2-weeks | 0.89 [0.82 to 10.36]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.191, Mixed Models Analysis

18. Primary Outcome: Change in IL-18 From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  IL-18 baseline 2-weeks | 9.61 [3.23 to 15.71]
  IL-18 last 2-weeks | 6.66 [2.99 to 13.61]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.088, Mixed Models Analysis

19. Primary Outcome: Change in IL-21 From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  IL-21 baseline 2-weeks | 29.96 [13.50 to 725.93]
  IL-21 last 2-weeks | 327.07 [27.30 to 644.85]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.478, Mixed Models Analysis

20. Primary Outcome: Change in IL-23 From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  IL-23 baseline 2-weeks | 0 [0 to 0]
  IL-23 last 2-weeks | 0 [0 to 0]

21. Primary Outcome: Change in IL-31 From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  IL-31 baseline 2-weeks | 0 [0 to 0]
  IL-31 last 2-weeks | 0 [0 to 0]

22. Primary Outcome: Change in IL-27 From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  IL-27 baseline 2-weeks | 86.51 [35.49 to 156.03]
  IL-27 last 2-weeks | 96.39 [74.66 to 126.15]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.016, Mixed Models Analysis

23. Primary Outcome: Change in LIF From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  LIF baseline 2-weeks | 4.93 [3.98 to 87.52]
  LIF last 2-weeks | 4.49 [4.19 to 84.25]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.025, Mixed Models Analysis

24. Primary Outcome: Change in G-CSF From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  G-CSF baseline 2-weeks | 37.78 [22.63 to 152.62]
  G-CSF last 2-weeks | 35.67 [23.26 to 146.67]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.012, Mixed Models Analysis

25. Primary Outcome: Change in GM-CSF From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  GM-CSF baseline 2-weeks | 5779.44 [3252.62 to 26170.25]
  GM-CSF last 2-weeks | 6377.62 [2456.04 to 29829.31]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.426, Mixed Models Analysis

26. Primary Outcome: Change in MIP-1α From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  MIP-1α baseline 2-weeks | 5.66 [2.85 to 63.75]
  MIP-1α last 2-weeks | 3.60 [2.33 to 56.10]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.042, Mixed Models Analysis

27. Primary Outcome: Change in SDF-1α From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  SDF-1α baseline 2-weeks | 148.14 [95.03 to 1886.42]
  SDF-1α last 2-weeks | 123.19 [98.62 to 1955.32]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.708, Mixed Models Analysis

28. Primary Outcome: Change in IP-10 From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  IP-10 baseline 2-weeks | 6.01 [4.59 to 8.50]
  IP-10 last 2-weeks | 5.28 [4.73 to 8.44]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.558, Mixed Models Analysis

29. Primary Outcome: Change in Eotaxin From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  eotaxin baseline 2-weeks | 36.54 [19.41 to 78.23]
  eotaxin last 2-weeks | 29.95 [22.0 to 80.96]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.350, Mixed Models Analysis

30. Primary Outcome: Change in RANTES From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  RANTES baseline 2-weeks | 57.00 [49.04 to 105.46]
  RANTES last 2-weeks | 57.27 [47.15 to 123.27]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.655, Mixed Models Analysis

31. Primary Outcome: Change in MIP-1β From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  MIP-1β baseline 2-weeks | 58.52 [18.91 to 288.14]
  MIP-1β last 2-weeks | 51.08 [35.79 to 272.44]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.248, Mixed Models Analysis

32. Primary Outcome: Change in MCP-1 From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  MCP-1 baseline 2-weeks | 24.30 [15.25 to 87.01]
  MCP-1 last 2-weeks | 25.38 [19.60 to 74.88]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.128, Mixed Models Analysis

33. Primary Outcome: Change in MCP-3 From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  MCP-3 baseline 2-weeks | 31.52 [22.67 to 80.02]
  MCP-3 last 2-weeks | 25.30 [17.96 to 81.00]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.065, Mixed Models Analysis

34. Primary Outcome: Change in MIG From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  MIG baseline 2-weeks | 47.81 [28.80 to 1480.33]
  MIG last 2-weeks | 35.98 [27.73 to 1520.40]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.962, Mixed Models Analysis

35. Primary Outcome: Change in TRAIL From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  TRAIL baseline 2-weeks | 23.42 [5.41 to 925.52]
  TRAIL last 2-weeks | 12.95 [7.42 to 975.70]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.402, Mixed Models Analysis

36. Primary Outcome: Change in CD40L From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  CD40L baseline 2-weeks | 41.97 [30.11 to 316.03]
  CD40L last 2-weeks | 35.78 [19.50 to 281.48]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.201, Mixed Models Analysis

37. Primary Outcome: Change in TGF-α From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  TGF-α baseline 2-weeks | 1.42 [0.53 to 2.75]
  TGF-α last 2-weeks | 0.58 [0.18 to 2.69]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.016, Mixed Models Analysis

38. Primary Outcome: Change in TGF-β From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  TGF-β baseline 2-weeks | 9.40 [7.03 to 159.01]
  TGF-β last 2-weeks | 7.80 [6.05 to 141.56]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.006, Mixed Models Analysis

39. Primary Outcome: Change in IFN-α From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  IFN-α baseline 2-weeks | 4.99 [3.19 to 16.76]
  IFN-α last 2-weeks | 4.15 [3.57 to 14.49]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.007, Mixed Models Analysis

40. Primary Outcome: Change in IFN-β From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  IFN-β baseline 2-weeks | 24.04 [14.07 to 215.46]
  IFN-β last 2-weeks | 19.10 [15.81 to 179.89]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.038, Mixed Models Analysis

41. Primary Outcome: Change in IFN-γ From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  IFN-γ baseline 2-weeks | 11.42 [5.99 to 31.35]
  IFN-γ last 2-weeks | 9.29 [7.18 to 25.99]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.032, Mixed Models Analysis

42. Primary Outcome: Change in TNF-α From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  TNF-α baseline 2-weeks | 124.36 [90.05 to 368.04]
  TNF-α last 2-weeks | 116.04 [89.75 to 339.64]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.002, Mixed Models Analysis

43. Primary Outcome: Change in TNF-β From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  TNF-β baseline 2-weeks | 0 [0 to 0]
  TNF-β last 2-weeks | 0 [0 to 0]

44. Primary Outcome: Change in PIGF-1 From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  PIGF-1 baseline 2-weeks | 1.75 [1.65 to 2.46]
  PIGF-1 last 2-weeks | 2.09 [1.98 to 2.40]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.508, Mixed Models Analysis

45. Primary Outcome: Change in SCF From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  SCF baseline 2-weeks | 7.53 [3.05 to 66.74]
  SCF last 2-weeks | 5.41 [2.21 to 65.39]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.119, Mixed Models Analysis

46. Primary Outcome: Change in HGF From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  HGF baseline 2-weeks | 187.27 [150.29 to 1627.38]
  HGF last 2-weeks | 189.33 [130.54 to 1582.27]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.326, Mixed Models Analysis

47. Primary Outcome: Change in VEGF-D From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  VEGF-D baseline 2-weeks | 2.62 [0.43 to 55.26]
  VEGF-D last 2-weeks | 3.30 [0.81 to 56.61]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.753, Mixed Models Analysis

48. Primary Outcome: Change in VEGF From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  VEGF baseline 2-weeks | 80.95 [29.94 to 710.36]
  VEGF last 2-weeks | 70.70 [33.64 to 689.66]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.067, Mixed Models Analysis

49. Primary Outcome: Change in NGF From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  NGF baseline 2-weeks | 12.24 [4.32 to 150.09]
  NGF last 2-weeks | 10.50 [1.88 to 139.01]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.080, Mixed Models Analysis

50. Primary Outcome: Change in EGF From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  EGF baseline 2-weeks | 5.23 [1.77 to 97.32]
  EGF last 2-weeks | 3.23 [0.35 to 41.64]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.639, Mixed Models Analysis

51. Primary Outcome: Change in FGF-β From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  FGF-β baseline 2-weeks | 0 [0 to 0]
  FGF-β last 2-weeks | 0 [0 to 0]

52. Primary Outcome: Change in M-CSF From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  M-CSF baseline 2-weeks | 0 [0 to 0]
  M-CSF last 2-weeks | 0 [0 to 0]

53. Primary Outcome: Change in BDNF From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  BDNF baseline 2-weeks | 777.60 [478.46 to 1687.16]
  BDNF last 2-weeks | 717.98 [399.81 to 1824.11]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.945, Mixed Models Analysis

54. Primary Outcome: Change in ICAM-1 From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  ICAM-1 baseline 2-weeks | 2670.81 [1368.85 to 4326.96]
  ICAM-1 last 2-weeks | 2820.63 [1569.72 to 3802.24]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.038, Mixed Models Analysis

55. Primary Outcome: Change in VCAM-1 From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  VCAM-1 baseline 2-weeks | 30876.40 [28221.23 to 54690.42]
  VCAM-1 last 2-weeks | 32156.99 [26838.15 to 70652.26]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.281, Mixed Models Analysis

56. Primary Outcome: Change in ENA-78 From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  ENA-78 baseline 2-weeks | 134.64 [20.40 to 226.86]
  ENA-78 last 2-weeks | 83.36 [16.32 to 197.58]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.030, Mixed Models Analysis

57. Primary Outcome: Change in PDGF-BB From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  PDGF-BB baseline 2-weeks | 179.89 [129.46 to 269.13]
  PDGF-BB last 2-weeks | 150.29 [122.19 to 305.54]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.948, Mixed Models Analysis

58. Primary Outcome: Change in PAI-1 From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  PAI-1 baseline 2-weeks | 15086.40 [13707.57 to 23919.29]
  PAI-1 last 2-weeks | 15536.99 [14295.96 to 29989.92]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.610, Mixed Models Analysis

59. Primary Outcome: Change in Leptin From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  leptin baseline 2-weeks | 3991.44 [1950.32 to 8616.49]
  leptin last 2-weeks | 4128.32 [1762.54 to 9120.73]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.893, Mixed Models Analysis

60. Primary Outcome: Change in Resistin From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  Resistin baseline 2-weeks | 1831.26 [1504.34 to 2771.75]
  Resistin last 2-weeks | 1942.47 [1722.55 to 3009.37]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.041, Mixed Models Analysis

61. Primary Outcome: Change in GROa From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  GROa baseline 2-weeks | 0 [0 to 0]
  GROa last 2-weeks | 0 [0 to 0]

62. Primary Outcome: Change in FaSL From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  FaSL baseline 2-weeks | 0 [0 to 0]
  FaSL last 2-weeks | 0 [0 to 0]

63. Primary Outcome: Change in IL-22 From Baseline.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
pg/mL
  IL-22 baseline 2-weeks | 194.59 [99.61 to 1193.80]
  IL-22 last 2-weeks | 220.62 [132.15 to 1012.50]
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p = 0.967, Mixed Models Analysis

64. Primary Outcome: Change in Pain From Baseline.
Description: Visual analog scale (0-100) anchored at "no pain" at 0 and "worst possible pain" at 100. Improvement in pain would be indicated by a decrease in the score.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
units on a scale
  Pain baseline 2-weeks | 51.149 (4.841)
  Pain last 2-weeks | 43.286 (4.805)
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p < 0.001, Mixed Models Analysis

65. Primary Outcome: Change in Overall Fibromyalgia Symptoms From Baseline.
Description: Visual analog scale (0-100) anchored at "no symptoms" at 0 and "worst possible symptoms" at 100. Improvement in overall fibromyalgia symptoms would be indicated by a decrease in the score.
Time Frame: Baseline period (2 weeks) through end of drug phase (8 weeks) [10 weeks total].
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Low Dose Naltrexone (LDN)
Number analyzed (Participants) | 8
units on a scale
  Overall symptoms baseline 2-weeks | 55.653 (4.671)
  Overall symptoms last 2-weeks | 45.506 (4.633)
Statistical Analysis 1: Comparison: Low Dose Naltrexone (LDN); Test type: Superiority or Other; p < 0.001, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 8 week drug administration period.
Arm/Group | Low Dose Naltrexone (LDN)
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

LIMITATIONS AND CAVEATS:
No placebo control drug used - participants were only advised that placebo may be used during the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes